CLINICAL TRIAL: NCT04569669
Title: A Clinical Trial on the Diagnostic Performance Based on CT-Derived Fractional Flow Reserve Score Analysis Software for Coronary Artery Stenosis
Brief Title: The Sensitivity and Specificity of CardioSimFFRct Analysis Software on Coronary Artery Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CCRF Inc., Beijing, China (Industry)
Collaborators: Shengshi Technology, Co., Ltd, Hangzhou, China (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SS-YF-101-LCF01-Z
Record Dates: First submitted 2020-07-30; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Coronary Stenosis
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients diagnosed with Coronary Artery Disease（CAD）by CCTA (Experimental): Patients admitted to hospital with the diagnosed of CAD by CCTA and who accept to participate to the study will undergo the invasive coronary angiography, fractional flow reserve (FFR) will be measured during the invasive coronary angiography.Outcome measures were comparing FFRct to FFR.
  Interventions: Diagnostic Test: FFR and FFRCT

INTERVENTIONS:
Diagnostic Test: FFR and FFRCT — All the patients will undergo computed coronary tomography angiography to analysis FFRCT . Then FFR will be measured during invasive cardiac catheterization.

SUMMARY:
The device involved in this trail is a diagnostic software with a Prospective, Multicenter, Self Controlled design. FFRCT diagnostic performance was calculated by CardioSimFFRct Analysis software, and the diagnostic accuracy, sensitivity, specificity, positive predictive value and negative predictive performance of FFRCT for myocardial ischemia were calculated per-patient level and per-vessel level with invasive FFR value as gold standard.

DETAILED DESCRIPTION:
The present study is a single arm, open label, prospective trial. Measurement of FFR during invasive cardiac catheterization represents the "gold standard" for assessment of the hemodynamic significance of coronary artery lesions. As we know, the major disadvantage of FFR is that it has to be measured invasively. CardioSimFFRct Analysis software is a non-invasive method to determine FFR which computes the hemodynamic significance of Coronary Artery Disease (FFRCT) from coronary computed tomography angiography（CCTA）data of the subject by using computational fluid dynamics.The FFR derived from FFR-CT will be compared with invasive FFR as gold standard.Moreover CardioSimFFRct also simplifies the coronary artery into a one-dimensional piping model, omits grid engineering, and greatly reduces the complexity of pretreatment.Based on the pressure loss along the pipe flow and the local pressure loss, a fast method for FFR calculation in engineering is proposed. The calculation time can be reduced to several minutes.

FFRct from CardioSimFFRct Analysis software is mainly based on CCTA images to image the coronary arteries. Through three-dimensional reconstruction of the coronary arteries and computational fluid Dynamics (CFD) technology, the simulation of blood flow in the blood vessels is realized to extract the coronary blood flow reserve score (FFR).FFRct has the following characteristics such as the FFR value can be measured noninvasively, without additional damage to patients, avoiding the risks brought by invasive surgery, and the side effects brought by drugs during invasive surgery.FFRct can realize the examination quickly, save the time of doctors' coronary functional assessment, and simplify the process of coronary functional assessment.It also has the function of three-dimensional reconstruction of blood vessels, which makes it convenient for users to view the whole structure of coronary arteries and make artificial correction.The results of FFRct have high repeatability and are easy for users to evaluate.

ELIGIBILITY:
Inclusion Criteria:

Subjects that participate in this study must fulfill all the following criteria:

General inclusion criteria:

* Age ≥18 years and ≤ 80 years;
* Subject providing written informed consent;
* After the researcher assessed the suspected presence of coronary artery stenosis, coronary angiography and CCTA examination were proposed.

Angiographic inclusion criteria:

* CCTA inspection should be performed on instruments with at least 64 multidetector rows;
* CCTA images are clear and readable;
* The diameter of coronary artery lesion stenosis was measured by CCTA image with 30%-90%;
* The reference vessel diameter of coronary stenosis was ≥2.5mm by CCTA imaging.

Exclusion Criteria:

If subjects fulfill any of below criteria, this subject shall be exclude from this study.

General exclusion criteria:

* Pregnant and breast-feeding women;
* Previous ST-segment elevation myocardial infarction 30 days before CCTA examination, and a history of non-ST-segment elevation myocardial infarction 7 days before CCTA examination;
* Prior Coronary Artery Bypass Graft（CABG）,Pacemaker, Implantable Cardioverter Defibrillator（ICD）, Artificial Valve Implantation;
* Hypertrophic obstructive cardiomyopathy;
* Heart failure(NYHA≥III or Left Ventricular Ejection Fraction（LVEF）< 40%);
* Atrial fibrillation, supraventricular tachycardia, ventricular tachycardia and other arrhythmias;
* Body mass index >35kg/m2;
* Serum creatinine >178µmol/L or 2mg/dl;
* Allergies or contraindications to contrast agents are known;
* Subject who received Nicorandil within 2 weeks prior to invasive FFR examination;
* Any other conditions that are not suitable for the study.

Angiographic exclusion criteria:

* The quality of CT imaging is not good enough to extract coronary blood vessel trees;
* Visual measurement of coronary lesion diameter stenosis > 90% by CCTA imaging;
* The target lesions were diffuse lesions, and the lesion length was ≥ 30mm (visual measurement);
* There were ≥ 2 stenosis lesions in the target vessel;
* Stent implantation in the target vessel;
* Lesions involving aneurysms or myocardial Bridges;
* The target vessel is very tortuous and it is difficult to predict the passage of the pressure guide wire.
* Left main disease;
* Patients with acute coronary syndrome after CCTA examination and before invasive FFR examination;
* Severe calcification(i.e Diffuse calcification ,Local or segmental calcification)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Estimated)
Dates: Start 2020-10-09 (Estimated); Primary Completion 2021-10-09 (Estimated); Study Completion 2022-03-09 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity (subject level) of FFRCT | Measurement at Procedure/Baseline Visit
  Sensitivity and specificity (subject level) for predicting the functional significance of coronary artery stenosis using CT-Derived Fractional Flow Reserve Score Analysis Software.

SECONDARY OUTCOMES:
AUC between FFRCT vs. FFR | Measurement at Procedure/Baseline Visit
  Comparing the Area Under Curve(AUC) between FFRct and CCTA to determine the Functional significance of coronary stenosis.
Sensitivity and Specificity between FFRCT vs. FFR | Measurement at Procedure/Baseline Visit
  Comparing the Sensitivity and Specificity which at the lesion level between FFRct and CCTA
Accuracy (lesion level and subject level) between FFRCT vs. FFR | Measurement at Procedure/Baseline Visit
  Comparing the Accuracy which at the lesion level and subject level between FFRct and CCTA
Positive Predictive Value (PPV) between FFRCT vs. FFR | Measurement at Procedure/Baseline Visit
  Comparing the positive predictive value (PPV) between FFRct and CCTA
Negative Predictive Value (NPV) between FFRCT vs. FFR | Measurement at Procedure/Baseline Visit
  Comparing the negative predictive value (NPV) between FFRct and CCTA

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, professor, Principal Investigator — The General Hospital of Northern Theater Command
Locations (8):
- China (8):
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Dalian University, Dalian, Liaoning
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - Tianjin Chest Hospital, Tianjing, Tianjing
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No